CLINICAL TRIAL: NCT04052165
Title: IOP Reduction and Complications of Polymethyl Methacrylate Glaucoma Drainage Device on Glaucoma Patient
Brief Title: IOP Reduction and Complications of Polymethyl Methacrylate GDD on Glaucoma Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Fakultas Kedokteran Universitas Indonesia (Other); Dr Cipto Mangunkusumo General Hospital (Other); Institut Pertanian Bogor (Other)
Responsible Party: Principal Investigator, Dr. dr. Virna Dwi Oktariana, SpM(K), Principal Investigator, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Oktariana
Record Dates: First submitted 2019-08-06; First posted 2019-08-09 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Glaucoma Eye
Keywords: Effectiveness; Glaucoma Drainage Device; Intraocular pressure; Tissue Response
MeSH Terms: interventions — Glaucoma Drainage Implants

STUDY DESIGN:
Intervention Model Description: GDD in glaucoma patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Glaucoma drainage device in glaucoma patient (Experimental): GDD is inserted in glaucoma patients
  Interventions: Procedure: Glaucoma Implant

INTERVENTIONS:
Procedure: Glaucoma Implant

SUMMARY:
Glaucoma is a group of diseases that damage the eye's optic nerve, result in progressive visual field defect and blindness. The aim of glaucoma management is to reduce IOP, and glaucoma implant surgery is the alternative treatment that can be chosen. The effectiveness of the implant on the end stage glaucoma patients was evaluated by the reduction of intra ocular pressure (IOP) and well formed blebs that were evaluated clinically and by using anterior scanning optical coherence tomography (AS-OCT). The safety of the implant was determined by the regression of the clinical symptoms and there were no severe complications such as implant extrusion. Two patients developed improvement of the visual acuity. This was an unpredictable positive result.

DETAILED DESCRIPTION:
The study is to measure the efficacy of new GDD that made with polymethyl methacrylate. The primary outcome is IOP reduction. The secondary outcome is glaucoma medication post surgery and complication that occurred during the follow up. The subjects are refractory glaucoma patients that need glaucoma drainage device implantation. The measurement are collected on first day, first month, third month, sixth month and twelve month. The IOP will be measured using GAT (Goldmann applanation tonometer), but if the subjects are not cooperative, they will be measured using i-care. On the follow up, the glaucoma medication needed will be noted and also for the complication and the need for other surgery, e.g. AC formation using viscoelastic, repair tube/plate exposure, cyclo photocoagulation, etc.

ELIGIBILITY:
Inclusion Criteria:

* End stage glaucoma patients whose IOP is failed to be controlled by glaucoma medications
* Patients that are willing to participate in the study
* Patients with <6/60 visual acuity
* Patients above 18 years

Exclusion Criteria:

* Patients with combination surgery indication (eg. glaucoma with cataracts)
* Eyes with congenital disease of anterior segment dysgenesis
* Eyes with uneven surface of the cornea that the measurement IOP with Goldmann tonometer could be difficult
* Eyes with broad conjungtival cicatrix that are impossible to be implanted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-08-08 (Actual)

PRIMARY OUTCOMES:
IOP reduction of Polymethylmethacrylate Glaucoma Drainage Device in refractory Glaucoma Patients | pre implantation surgery, day 1, 7, 30, 60, 90 post implantation surgery
  Intraocular pressure (IOP)

SECONDARY OUTCOMES:
The glaucoma medication that was used pre and post operative | pre implantation surgery, day 1, 7, 30, 60, 90 post implantation surgery
  The glaucoma medication used pre and post op
The complications that occurred during the follow up | during the surgery, day 1, 7, 30, 60, 90 post implantation surgery
  The complications that occurred during the follow up

CONTACTS AND LOCATIONS:
Overall Officials: Virna Dwi Oktariana Asrory, PhD, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giangiacomo A, Coleman AL. The Epidemiology of Glaucoma. In: Grehn F, Stamper R, editors. Glaucoma [Internet]. Berlin, Heidelberg: Springer Berlin Heidelberg; 2009 [cited 2016 Jun 14]. p. 13-21. Available from: http://link.springer.com/10.1007/978-3-540-69475-5_2
- [Background] Stamper R, Lieberman M, Drake M. Introduction and Classification of the Glaucomas. In: Becker-Shaffer's Diagnosis and Therapy of the Glaucomas. 8th ed. Mosby Elsevier; 2009. p. 1-7.
- [Background] Stamper R, Drake M, Lieberman M. Primary Open Angle Glaucoma. In: Becker-Shaffer's Diagnosis and Therapy of the Glaucomas. 8th ed. Mosby Elsevier; 2009. p. 239-57
- [Background] Sharaawy T, Sherwood M, Hitchings R. Glaucoma. 1st ed. Vol. 1. Philadelphia: Saunder Elsevier; 2009.
- [Background] Stamper RL, Lieberman MF, Drake MV. Laser Therapy. In: Becker-Shaffer's Diagnosis and Therapy of the Glaucomas. 8th ed. USA: Elsevier Health Sciences; 2009. p. 436-8.
- [Background] Stamper RL, Lieberman MF, Drake MV. Glaucoma outflow procedure. In: Becker-Shaffer's Diagnosis and Therapy of the Glaucomas. UK: Elsevier Health Sciences; 2009. p. 466-90.
- [Background] Eisenberg DL, Koo EY, Hafner G, Schuman JS. In vitro flow properties of glaucoma implant devices. Ophthalmic Surg Lasers. 1999 Sep-Oct;30(8):662-7. PMID 10507569
- [Background] Koura Y, Fukushima A, Nishino K, Ishida W, Nakakuki T, Sento M, Yamazoe K, Yamaguchi T, Misyoshi T, Ueno H. Inflammatory reaction following cataract surgery and implantation of acrylic intraocular lens in rabbits with endotoxin-induced uveitis. Eye (Lond). 2006 May;20(5):606-10. doi: 10.1038/sj.eye.6701975. PMID 15999134
- [Background] Kim MS, Rhee SW. Effects on the surrounding tissues and morphological changes of components after implantation of PMMA and heparin surface modified PMMA intraocular lens in rabbit eyes. Korean J Ophthalmol. 1990 Dec;4(2):73-81. doi: 10.3341/kjo.1990.4.2.73. PMID 2092164
- [Background] Cioffi G. Basic and Clinical Science Course. 11th ed. American Academy of Ophtalmology; 2011. 211-215 p.
- [Background] Wilson MR, Mendis U, Smith SD, Paliwal A. Ahmed glaucoma valve implant vs trabeculectomy in the surgical treatment of glaucoma: a randomized clinical trial. Am J Ophthalmol. 2000 Sep;130(3):267-73. doi: 10.1016/s0002-9394(00)00473-6. PMID 11020403
- [Background] Beck AD, Freedman S, Kammer J, Jin J. Aqueous shunt devices compared with trabeculectomy with Mitomycin-C for children in the first two years of life. Am J Ophthalmol. 2003 Dec;136(6):994-1000. doi: 10.1016/s0002-9394(03)00714-1. PMID 14644208
- [Background] Jung KI, Lim SA, Park HY, Park CK. Visualization of blebs using anterior-segment optical coherence tomography after glaucoma drainage implant surgery. Ophthalmology. 2013 May;120(5):978-83. doi: 10.1016/j.ophtha.2012.10.015. Epub 2013 Jan 21. PMID 23347982
- [Background] Azuara-Blanco A, Katz LJ. Dysfunctional filtering blebs. Surv Ophthalmol. 1998 Sep-Oct;43(2):93-126. doi: 10.1016/s0039-6257(98)00025-3. PMID 9763136
- [Background] Clark A, Wax M, Civan M. Mechanisms of Glaucoma. In: Ophthalmology. 3rd ed. St. Louis, Mo: Mosby Elsevier; 2014. p. 1012-8.
- [Background] Chang DT, Jones JA, Meyerson H, Colton E, Kwon IK, Matsuda T, Anderson JM. Lymphocyte/macrophage interactions: biomaterial surface-dependent cytokine, chemokine, and matrix protein production. J Biomed Mater Res A. 2008 Dec 1;87(3):676-87. doi: 10.1002/jbm.a.31630. PMID 18200554
- [Background] Major MR, Wong VW, Nelson ER, Longaker MT, Gurtner GC. The foreign body response: at the interface of surgery and bioengineering. Plast Reconstr Surg. 2015 May;135(5):1489-1498. doi: 10.1097/PRS.0000000000001193. PMID 25919260